CLINICAL TRIAL: NCT05949268
Title: Video Capsule Endoscopy for Detection of Gastrointestinal Bleeding in the Jejunum
Brief Title: Video Capsule Endoscopy for Detection of Gastrointestinal Bleeding in the Small Bowel
Status: Recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dominik Bettinger, Principal Investigator, University Hospital Freiburg
Other Study IDs: Capsule endoscopy_FR
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: GastroIntestinal Bleeding
Keywords: Small bowel capsule endoscopy; gastrointestinal bleeding; anticaogulation
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with gastrointestinal bleeding undetected in gastroscopy and colonoscopy: Gastrointestinal bleeding in the small bowel.
  Interventions: Device: Small bowel capsule endoscopy

INTERVENTIONS:
Device: Small bowel capsule endoscopy — Patients with gastrointestinal bleeding receive small bowel capsule endoscopy after bleeding could not be located in gastroscopy or colonoscopy.

SUMMARY:
Small bowel capsule endoscopy is the main diagnostic standard for small bowel bleeding. This study investigates the detection rate of small bowel bleeding in capsule endoscopy and further endoscopic treatment in a prospective and retrospective cohort.

DETAILED DESCRIPTION:
Small bowel capsule endoscopy is considered the diagnostic gold standard in the diagnosis of diseases of the small bowel. Most indications for capsule endoscopy are overt small bowel bleedings - defined as gastrointestinal bleeding after negative gastroscopy and colonoscopy - or occult iron deficiency anemia. Timing of small bowel capsule endoscopy seems to be decisive for the diagnosis of small bowel bleeding: corresponding to the actual guidelines the detection of small bowel bleeding can be up to > 70% if the intervention is performed within 2 days. Treatment of small bowel bleedings can be performed with small bowel enteroscopy such as balloon or motorized spiral enteroscopy. Against this background this study investigates the rate of small bowel bleeding diagnosed in capsule endoscopy. The aim of the study is to report tumorous, vascular and inflammatory findings as well as complications and cecal accessibility. One focus of the study is the time between small bowel bleeding and small bowel capsule endoscopy and small bowel enteroscopy, respectively. Endoscopic therapies and further bleeding episodes are recorded. In order to determine the improved clinical outcome after the introduction of the shortened timing for recommendation published in 2022, a retrospective cohort should be included in addition to a prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of gastrointestinal bleeding in the small bowel undetected by gastroscopy and colonoscopy
* informed consent

Exclusion Criteria:

* contraindications for small bowel capsule endoscopy (e.g. stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present with gastrointestinal bleeding undetected in gastroscopy or colonoscopy will be included in this cohort study. In these patients bleeding in the small bowel is suspected and they are allocated to a diagnostic assessment with small bowel capsule endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of small bowel bleeding detected during small bowel capsule endoscopy | Through study completion, an average of 1 year
  Detection of bleeding during small bowel capsule endoscopy

SECONDARY OUTCOMES:
Prevalence of vascular lesions as source of bleeding | Through study completion, an average of 1 year
  Detection of vascular lesions angiodysplasia) as source of bleeding
Prevalence of inflammatory lesions as source of bleeding | Through study completion, an average of 1 year
  Detection of inflammatory lesions as source of bleeding
Prevalence of tumor lesions as source of bleeding | Through study completion, an average of 1 year
  Detection of tumor lesions as source of bleeding
Complications of small bowel capsule endoscopy | Through study completion, an average of 1 year
  Complications of small bowel capsule endoscopy
Technical success of small bowel capsule endoscopy | Through study completion, an average of 1 year
  Technical success is defined as arrival of the capsule in the cecum
Time between diagnostic small bowel capsule endoscopy and small bowel enteroscopy for treatment of bleeding | From time to the end of capsule endoscopy until beginning of small bowel enteroscopy
  Time between diagnostic mall bowel capsule endoscopy and small bowel enteroscopy for treatment of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schultheiss, MD, Principal Investigator — University Medical Center Freiburg, Department of Medicine II, Freiburg, Germany
Locations (1):
- University Medical Center Freiburg, Department of Medicine II, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No
IPD are shared on reasonable request to the Principal Investigator.

REFERENCES:
- [Background] Rondonotti E, Spada C, Adler S, May A, Despott EJ, Koulaouzidis A, Panter S, Domagk D, Fernandez-Urien I, Rahmi G, Riccioni ME, van Hooft JE, Hassan C, Pennazio M. Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Technical Review. Endoscopy. 2018 Apr;50(4):423-446. doi: 10.1055/a-0576-0566. Epub 2018 Mar 14. PMID 29539652